CLINICAL TRIAL: NCT03453372
Title: Pain in Knee Osteoarthritis, a Placebo-controlled Randomized Clinical Trial for a New Potential Therapeutic Approach: Magnetic Resonance Guided Focused Ultrasound Surgery (MRgFUS)
Brief Title: MRgFUS in the Treatment of Osteoarthritic Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: knee@IORFus
Record Dates: First submitted 2018-02-23; First posted 2018-03-05 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-03

CONDITIONS: Osteo Arthritis Knee; Osteoarthritis; Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee; MRgFUS; ExAblate; Pain; High-Intensity Focused Ultrasound Ablation
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Pain

STUDY DESIGN:
Intervention Model Description: Double-blind placebo-controlled randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: Participating patients will be blinded to treatment assignment and to the ongoing results of the study; they will remain blinded to their assignment throughout the study period. All the staff involved in the pre- and post-treatment evaluation of patients will be also blinded. The evaluation of patients will be performed by physicians not involved in the treatment to ensure double blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental): MRgFUS treatment of pain caused by knee osteoarthritis
  Interventions: Device: MRgFUS Treatment
- Placebo (Placebo Comparator): Procedures in the placebo group will be identical to procedures in the active group, except no sonications (ultrasound emission) will be used.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: MRgFUS Treatment — Treatment of pain caused by knee osteoarthritis with high-intensity focused ultrasound
  Arms: Active
Other: Placebo — Procedures in the placebo group will be identical to procedures in the active group, except no sonications (ultrasound emission) will be used.
  Arms: Placebo

SUMMARY:
A double-blind placebo-controlled randomized clinical trial to evaluate the efficacy of magnetic resonance-guided focused ultrasound surgery (MRgFUS) in the treatment of pain caused by knee osteoarthritis (OA)

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a common, disabling, and costly disease, and the knee is one of the most affected joints. The predominant symptom is pain. Effective and lasting non-invasive treatment approaches are missing. MR-guided focused ultrasound surgery (MRgFUS) is a new minimally invasive technique which may represent a valid solution providing several advantages. The primary aim of this work will be to assess the efficacy of MRgFUS in the treatment of pain caused by knee OA in 80 patients candidate for arthroplasty in a prospective, randomized, double-blinded, placebo-controlled clinical trial. Different parameters related to pain, quality of life, function, and imaging will be collected and analyzed in a 12-month follow-up. The secondary aims will be focused on a) the evaluation of the effects on the joint organ and changes of biological features in response to MRgFUS, and b) the impact of selective ablation of nociceptors on OA pain, based on the analysis of resected joint tissues.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 50-80 years
* Activity-related joint pain
* Patients who have not responded to previous treatments and patients candidate for surgery
* Kellgren-Lawrence score 2-4 on X-rays
* Patients able to give their informed consent

Exclusion Criteria:

* Prior surgery in the past 12 months or previous local treatment in the past 3 months
* Changes in medications used during the previous 2 months
* Corticosteroid use for more than 3 months within the preceding year
* Rheumatologic and neurological disorders
* Fibromyalgia
* Trauma, fracture or osteomyelitis of the investigated joints within the preceding year
* Pregnancy
* Patients with large scars potentially included in the ultrasound beam path
* General contraindications to MRI and/or to anaesthesiological procedures
* Presence of internal hardware or device potentially affecting MR thermometry
* Patients involved in other clinical studies

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2020-01-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of MRgFUS in the treatment of pain caused by knee OA | Baseline (Day 1), 24 hours post MRgFUS, Week 1, 2, 3, Month 1, 3, 6,12
  The efficacy of MRgFUS will be demonstrated if the treatment group has a mean reduction of Visual Analog Pain Scale (VAS) of at least 1.5 points greater than the control group.

SECONDARY OUTCOMES:
Effects of MRgFUS on the joint organ: inflammation | Baseline (Day 1), 24 hours post MRgFUS, Month 1, 3, 6,12
  Enzyme linked immuno assays kits will be used to test inflammatory markers in serum. The reference standard values of the standardized markers will be considered for the evaluations.
Effects of MRgFUS on the joint organ: bone turnover | Baseline (Day 1), 24 hours post MRgFUS, Month 1, 3, 6,12
  Enzyme linked immuno assays kits will be used to test bone turnover markers in serum. The reference standard values of the standardized markers will be considered for the evaluations.
Effects of MRgFUS on the joint organ: pain | Baseline (Day 1), 24 hours post MRgFUS, Month 1, 3, 6,12
  Enzyme linked immuno assays kits will be used to test pain markers in serum. The reference standard values of the standardized markers will be considered for the evaluations.
Effects of MRgFUS on the joint organ: cartilage turnover | Baseline (Day 1), 24 hours post MRgFUS, Month 1, 3, 6,12
  Enzyme linked immuno assays kits will be used to test cartilage turnover markers in urine. The reference standard values of the standardized markers will be considered for the evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Bazzocchi, MD, PhD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided